CLINICAL TRIAL: NCT02656797
Title: Topical Liposomal Amphotericin B Gel Treatment for Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, AMIR HOREV, Head, Pediatric dermatology Service, Soroka University Medical Center, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sor017715ctil
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Leishmaniasis
Keywords: Leishmania major; Leishmania tropica; Amphotericin B
MeSH Terms: conditions — Leishmaniasis | interventions — Amphotericin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AM-B (Experimental): Topical Amphotericin-B 0.4% liposomal gel
  Interventions: Drug: Topical Amphotericin-B 0.4% liposomal gel
- Placebo (Placebo Comparator): Placebo gel preparation
  Interventions: Drug: Topical Amphotericin-B 0.4% liposomal gel

INTERVENTIONS:
Drug: Topical Amphotericin-B 0.4% liposomal gel — Topical Amphotericin-B 0.4% liposomal gel

SUMMARY:
Comparison between placebo gel treatment to topical liposomal amphotericin B gel treatment for cutaneous leishmaniasis of Leishmania species major and tropica.

DETAILED DESCRIPTION:
Randomized, double blind, placebo controlled study. The study will include 108 patients with cutenous leishmaniasis of Leishmania species major and tropica, confired by Polymerase Chain Reaction of a sample from a lesion.

Cure rate will be compared between patients treated with Amphotericin-B 0.4% Liposomal Gel and patients treated with placebo gel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Cutenous leishmaniasis confirmed by PCR (Leishmania species major or tropica)
* 1 to 5 lesions
* Signed informed consent

Exclusion Criteria:

* Facial lesions
* Significant co-morbidity
* Pregnancy or breast-feeding at enrollment
* Previous treatment for leishmaniasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Complete re-epithelization | Day 28 from enrollement
  Absence of ulceration, induration, erosion and

SECONDARY OUTCOMES:
Lesion size | Day 28 and day 56 from enrollement
  Defined by the multiplication of lesion length and width
Complete re-epithelization | Day 28 from enrollement
Skin manifestations | Day 28 and day 56 from enrollement
  Pruritus, pain, etching, discharge, bloating
Evidence of lesihmania infection | Day 56 from enrollement
  Evaluated by PCR test from a sample acquired from the lesion

CONTACTS AND LOCATIONS:
Overall Officials: Amir Horev, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No